CLINICAL TRIAL: NCT06214819
Title: Randomized, Controlled, Open-label, Double-blind, Multicenter Investigation Plan to Evaluate Early Endothelialization of a Polymer Free Sirolimus-eluting Coronary Stent System (VIVO ISARTM) Compared With Everolimus-eluting Durable Polymer Stent (XIENCE SkypointTM) in Patients Undergoing Percutaneous Coronary Intervention.
Brief Title: Plan to Evaluate Early Endothelialization of a Polymer Free Sirolimus-eluting Coronary Stent System (VIVO ISARTM) Compared With Everolimus-eluting Durable Polymer Stent (XIENCE SkypointTM) in Patients Undergoing Percutaneous Coronary Intervention.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC31-PRO-HEAL TRIAL
Record Dates: First submitted 2023-12-13; First posted 2024-01-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stents; Strut coverage by optic coherence tomography; Early endothelization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIVO ISAR DES in the first lesion (Experimental)
  Interventions: Device: VIVO ISAR DES implanted in the First lesion, XIENCE Skypoint DES implanted in the Second lesion
- XIENCE Skypoint DES in the first lesion (Active Comparator)
  Interventions: Device: XIENCE Skypoint DES implanted in the First lesion, VIVO ISAR DES implanted in the Second lesion

INTERVENTIONS:
Device: VIVO ISAR DES implanted in the First lesion, XIENCE Skypoint DES implanted in the Second lesion — VIVO ISAR DES implanted in the First lesion, XIENCE Skypoint DES implanted in the Second lesion
  Arms: VIVO ISAR DES in the first lesion
Device: XIENCE Skypoint DES implanted in the First lesion, VIVO ISAR DES implanted in the Second lesion — XIENCE Skypoint DES implanted in the First lesion, VIVO ISAR DES implanted in the Second lesion
  Arms: XIENCE Skypoint DES in the first lesion

SUMMARY:
To evaluate the stent endothelialization (> 20 microns) of VIVO ISARTM versus XIENCE SkypointTM stents at 1-month (very early strut covered) at follow-up by Optical Coherence Tomography (OCT) implanted IN THE SAME PATIENT during routine clinical practice.

DETAILED DESCRIPTION:
To evaluate the stent endothelialization (> 20 microns) of VIVO ISARTM versus XIENCE SkypointTM stents at 1-month (very early strut covered) at follow-up by Optical Coherence Tomography (OCT) implanted IN THE SAME PATIENT during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 18 years AND
* Patients who have signed informed consent AND
* Patients with coronary artery disease requiring percutaneous treatment with coronary stents due to de novo lesions in vessels with a diameter of reference from 2.25 mm to 4.0 mm AND
* Patients with at least 2 angiographic lesions in 2 different major coronary arteries. Or in the main branch and in one of its subsidiaries branches , as long as those are not "downstream" of the lesion from the main branch

Exclusion Criteria:

* Express refusal of the patient to participate in the study
* Patients with ST elevation Myocardial Infarction or Cardiogenic Shock
* Patients with high thrombotic content
* Pregnant or breastfeeding patients
* Patients with complex PCI (Percutaneous Coronary Intervention )(defined as):

  * Left main PC
  * Chronic total PC occlusion
  * Bifurcation lesion requiring 2-stent technique .
* Severe calcified lesion (need to use prior complex techniques of calcium modification such as intravascular lithotripsy, rotational/orbital atherectomy, laser.
* Patients with malignant neoplasms or other comorbid conditions with life expectancy <12 months
* Patients with a target lesion in a bypass graft
* Lesions due to restenosis
* Patients with PCI in the target vessel in the previous 9 months
* Patients with contraindication or difficulty to evaluate in the follow-up with OCT (renal failure, excessive tortuosity or lesions aorto-ostial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of early Covered struts (≥ 20μm) at 1 month OCT after stent implantation | 1 month
  Percentage of early Covered struts (≥ 20μm) at 1 month OCT after stent implantation
Percentage of stents with uncovered struts at 1 month OCT after stent implantation | 1 month
  Percentage of stents with uncovered struts (0μm) at 1 month OCT after stent implantation
Mean thickness of struts tissue coverage at 1 month OCT after stent implantation | 1 month
  Mean thickness of struts tissue coverage at 1 month OCT after stent implantation

SECONDARY OUTCOMES:
Percentage of malapposition of stent at 1 month OCT after stent implantation | 1 month
  Percentage of malapposition of stent at 1 month OCT after stent implantation
Percentage of covered struts at 1 months OCT after stent implantation | 1 month
  Percentage of covered struts at 1 months OCT after stent implantation
All-Cause Death Rate at 6 months | 6 months
  All-Cause Death Rate at 6 months
Cardiac Death Rate at 6 months | 6 months
  Cardiac Death Rate at 6 months
Myocardial Infarction Rate at 6 months | 6 months
  Myocardial Infarction Rate at 6 months
Target vessel revascularization Rate at 6 months | 6 months
  Target vessel revascularization Rate at 6 months
Neointimal Healing Score (NHC) by OCT at 1 month | 1 months
  The NHS is then calculated as follows:
  1. Presence of filling defect (% intraluminal defect, ILD) is assigned a weight of "4"
  2. Presence of both malapposed and uncovered struts (% malapposed/uncovered, MU) is assigned a weight of "3"
  3. Presence of uncovered struts alone (% malapposed, M) is assigned a weight of "2"
  4. Presence of malapposed struts alone (% uncovered, U) is assigned a weight of "1" Neointimal healing score = (%ILD * 4)+(%MU * 3)+(%U * 2)+(%M * 1).
Percentage of malapposed total struts at 1 month | 1 month
  Percentage of malapposed total struts at 1 month
Percentage of malapposed scaffold struts over side branch at 1 month | 1 month
  Strut malapposition: Measured maximum distance ≥100 μm between the strut surface and adjacent vessel surface by OCT, considering thickness of scaffold, was defined as malapposition. As a result, scaffold malapposition is defined as the presence of any malapposed struts. The ratio of malapposed struts (% malapposed strut) was the ratio of malapposed struts from total analyzable struts.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario de Gerona Doctor Josep Trueta, Girona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat

REFERENCES:
- [Background] Koppara T, Tada T, Xhepa E, Kufner S, Byrne RA, Ibrahim T, Laugwitz KL, Kastrati A, Joner M. Randomised comparison of vascular response to biodegradable polymer sirolimus eluting and permanent polymer everolimus eluting stents: An optical coherence tomography study. Int J Cardiol. 2018 May 1;258:42-49. doi: 10.1016/j.ijcard.2018.01.011. PMID 29544956
- [Background] Asano T, Jin Q, Katagiri Y, Kogame N, Takahashi K, Chang CC, Chichareon P, Wang C, Shi B, Su X, Fu G, Wu Y, Zhou X, Yuan Z, Wykrzykowska JJ, Piek JJ, Serruys PW, Onuma Y, Chen Y. A randomised comparison of healing response between the BuMA Supreme stent and the XIENCE stent at one-month and two-month follow-up: PIONEER-II OCT randomised controlled trial. EuroIntervention. 2018 Dec 20;14(12):e1306-e1315. doi: 10.4244/EIJ-D-18-00461. PMID 30082261
- [Background] Andreasen LN, Balleby IR, Barkholt TO, Hebsgaard L, Terkelsen CJ, Holck EN, Jensen LO, Maeng M, Dijkstra J, Antonsen L, Kristensen SD, Tu S, Lassen JF, Christiansen EH, Holm NR. Early healing after treatment of coronary lesions by thin strut everolimus, or thicker strut biolimus eluting bioabsorbable polymer stents: The SORT-OUT VIII OCT study. Catheter Cardiovasc Interv. 2023 Mar;101(4):787-797. doi: 10.1002/ccd.30579. Epub 2023 Feb 5. PMID 36740229
- [Background] Otaegui Irurueta I, Gonzalez Sucarrats S, Barron Molina JL, Perez de Prado A, Massotti M, Carmona Ramirez MA, Marti G, Bellera N, Serra B, Serra V, Domingo E, Lopez-Benito M, Sabate M, Ferreira Gonzalez I, Garcia Del Blanco B. Can an ultrathin strut stent design and a polymer free, proendothelializing probucol matrix coating improve early strut healing? The FRIENDLY-OCT trial. An intra-patient randomized study with OCT, evaluating early strut coverage of a novel probucol coated polymer-free and ultra-thin strut sirolimus-eluting stent compared to a biodegradable polymer sirolimus-eluting stent. Int J Cardiol. 2022 Aug 1;360:13-20. doi: 10.1016/j.ijcard.2022.04.043. Epub 2022 Apr 25. PMID 35472561
- [Background] Massberg S, Byrne RA, Kastrati A, Schulz S, Pache J, Hausleiter J, et al. Polymerfree sirolimus- and probucol-eluting versus new generation zotarolimus-eluting stents in coronary artery disease: the Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting versus Zotarolimus-eluting Stents (ISARTEST 5) trial. Circulation. 2 de agosto de 2011;124(5):624-32. 18. Kufner S, Sorges J, Mehilli J, Cassese S, Repp J, Wiebe J, et al. Randomized Trial of Polymer-Free Sirolimus- and Probucol-Eluting Stents Versus Durable Polymer Zotarolimus-Eluting Stents: 5-Year Results of the ISAR-TEST-5 Trial. JACC Cardiovasc Interv. 25 de abril de 2016;9(8):784-92.